CLINICAL TRIAL: NCT02389673
Title: Intra-operative Radiotherapy After Breast-conversing Surgery in Treating Women With Ductal Carcinoma in Situ Breast Cancer
Brief Title: Intra-operative Radiotherapy For Women With Ductal Carcinoma in Situ Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liao Ning (Other)
Responsible Party: Sponsor-Investigator, Liao Ning, Guangdong Academy of Medical Sciences, Guangdong Academy of Medical Sciences
Organization: Guangdong Academy of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGHBCRG-IORT-DCIS
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Breast Neoplasms
Keywords: Intermediate and high grade ductal carcinoma in situ （DCIS）
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Without Radiotherapy (No Intervention): Patients just accept breast-conversing surgery without radiotherapy.
- Intraoperative Radiotherapy (Experimental): Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  Interventions: Device: Intraoperative Radiotherapy

INTERVENTIONS:
Device: Intraoperative Radiotherapy — Boost with 20 Gy during BCS, EBRT with 46-50 Gy
  Arms: Intraoperative Radiotherapy

SUMMARY:
Whether the patients with low grade ductal carcinoma in situ breast cancer should accept radiationtherapy is uncertain.Radiation therapy uses high-energy x-rays to damage tumor cells. Giving radiation during surgery followed by external-beam radiation to the entire breast may kill more tumor cells.The clinical trial is conducting to find out the effectiveness of radiation therapy during surgery in treating women who have undergone breast-conversing surgery for low grade ductal carcinoma in situ breast cancer.

DETAILED DESCRIPTION:
Giving radiation during surgery followed by external-beam radiation to the entire breast may kill more tumor cells.The clinical trial is conducting to find out the effectiveness of radiation therapy during surgery in treating women who have undergone breast-conversing surgery for low grade ductal carcinoma in situ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Tumor diameter < 5 cm
* Low grade ductal carcinoma in situ
* Candidate for breast-conserving surgery
* Must have undergone lumpectomy with negative margins or minimal margin involvement
* Currently undergoing re-excision of the biopsy cavity and/or sentinel lymph node biopsy or axillary lymph node dissection
* No evidence of metastatic disease
* Informed consent

Exclusion Criteria:

* No informed consent
* Tumor size > 5 cm
* Intermediate or high grade ductal carcinoma in situ
* Invasive carcinoma
* No indication for a boost

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2014-10; Primary Completion 2019-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
ipsilateral breast tumor recurrence rate after surgery within five years | Within 5 years after surgery
  Within 5 years after surgery,we should evaluate ipsilateral breast tumor recurrence and Disease free survival as the most important outcome measure

SECONDARY OUTCOMES:
Disease free survival after surgery within five years | Within 5 years after surgery
  Within 5 years after adjuvant chemotherapy,we should evaluateDisease free survival(DFS) rates as thet important outcome measure.
Overall survival after surgery within ten years | Within ten years after surgery
  After surgery,we should evaluate overall survival (OR)rates as the secondary important outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Ning, MD,PhD, Study Director — Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China